CLINICAL TRIAL: NCT01797783
Title: Clinical Evaluation of the Safety and Efficacy of a New Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-12-054
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-04

CONDITIONS: Myopia; Ametropia; Presbyopia; Refractive Error
Keywords: Myopia; Presbyopia; Refractive error; Contact lenses; Multifocal
MeSH Terms: conditions — Myopia; Refractive Errors; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAILIES® AquaComfort Plus® Multifocal (Experimental): Nelfilcon A multifocal contact lens with comfort additive worn for 30 days on a daily wear, daily disposable basis
  Interventions: Device: Nelfilcon A multifocal contact lens with comfort additive
- Focus® DAILIES® Progressives (Active Comparator): Nelfilcon A multifocal contact lens worn for 30 days on a daily wear, daily disposable basis
  Interventions: Device: Nelfilcon A multifocal contact lens

INTERVENTIONS:
Device: Nelfilcon A multifocal contact lens with comfort additive
  Arms: DAILIES® AquaComfort Plus® Multifocal
Device: Nelfilcon A multifocal contact lens
  Arms: Focus® DAILIES® Progressives

SUMMARY:
The purpose of this study was to demonstrate substantial equivalence of the new DAILIES® AquaComfort Plus® Multifocal (DACP MF) contact lens to the commercially available Focus® DAILIES® Progressives (FDP) contact lens.

ELIGIBILITY:
Inclusion Criteria:

* Sign Informed Consent Document.
* Presbyopic and require a spectacle add of up to and including 3.00 diopters (D).
* Currently wear soft contact lenses.
* Willing and able to wear multifocal contact lenses in both eyes within the available range of powers for this trial and comply with the wearing and replacement schedule.
* Manifest cylinder less than or equal to 1.00 D.
* Able to achieve best corrected visual acuity (BCVA) of 20/25 or better (Snellen) in each eye at distance (as determined by manifest refraction).
* Able to achieve distance visual acuity of 20/40 (Snellen) or better in each eye with study lenses and deem subjective vision as satisfactory at time of dispense.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear within 6 months prior to enrollment.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated.
* History of corneal or refractive surgery.
* Biomicroscopy findings greater than Grade 2 at baseline.
* A pathologically dry eye that precludes contact lens wear.
* Monocular (only one eye with functional vision).
* Wear habitual contact lenses on an extended wear schedule (any number of nights of overnight wear on a regular basis).
* History of intolerance or hypersensitivity to any component of the investigational products.
* Concurrent participation in a contact lens or contact lens care product clinical trial or within the previous 30 days.
* Eye injury or ocular or intra-ocular surgery within 6 months prior to enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Webb, O.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 9 study centers located in the United States.
Pre-assignment Details: Of the 83 consented participants, 2 were exited as screen failures prior to randomization, and 2 were exited after randomization but prior to product dispense. This reporting group includes all randomized participants who were dispensed study product (79).
Period: Overall Study
Arm/Group | DAILIES® AquaComfort Plus® Multifocal | Focus® DAILIES® Progressives
Started | 52 | 27
Completed | 50 | 26
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants who were dispensed study product (79).
Groups:
- Total: Total of all reporting groups
Arm/Group | DAILIES® AquaComfort Plus® Multifocal | Focus® DAILIES® Progressives | Total
Number analyzed (Participants) | 52 | 27 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (5.19) | 49.7 (5.21) | 49.8 (5.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 22 | 56
  Male | 18 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Vision
Description: The participant was instructed to, "Please rate the aggregate of distance, intermediate, and near vision quality. Fill in the circle below the number that indicates your selection. Rate eyes together, marking only 1 circle for both eyes. Higher numbers mean better vision." The response was recorded on a continuous scale from 1-10 (1=poor, 10=excellent).
Time Frame: Up to Day 30
Population: This analysis population includes all randomized and dispensed participants who completed the study. No imputation was used for missing values. Here, "n" is the number of participants with non-missing values at the specific time point for each arm.
  group,
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus® Multifocal | Focus® DAILIES® Progressives
Number analyzed (Participants) | 50 | 26
Units on a scale
  Dispense (Day 0) (n=49,26) | 8.7 (1.1) | 8.4 (1.2)
  Day 3 (n=49,26) | 8.4 (1.3) | 7.5 (1.7)
  Day 14 (n=50,26) | 8.6 (1.2) | 7.7 (1.9)
  Day 30 (n=50,26) | 8.5 (1.1) | 7.6 (1.9)

2. Secondary Outcome: Binocular Snellen Visual Acuity (VA) at Distance With Study Lenses
Description: Visual Acuity was tested while reading a chart at 20-foot equivalent distance from the participant with both eyes together. The Snellen fraction compares the participant's result to the result expected from the 'normal' visual system. The numerator represents the distance between the participant and the chart, and the denominator represents the distance at which a person with 'normal' vision would be able to discern the same letter size. 20/20 is considered to be 'normal' vision, whereas visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity.
Time Frame: Up to Day 30
Population: This analysis population includes all randomized and dispensed participants who completed the study.
Measure: Number; unit: participants
Groups:
- DACP MF @ Dispense; DACP MF @ Day 3; DACP MF @ Day 14; DACP MF @ Day 30: Nelfilcon A multifocal contact lens with comfort additive worn for 30 days on a daily wear, daily disposable basis
- FDP @ Dispense; FDP @ Day 3; FDP @ Day 14; FDP @ Day 30: Nelfilcon A multifocal contact lens worn for 30 days on a daily wear, daily disposable basis
Arm/Group | DACP MF @ Dispense | DACP MF @ Day 3 | DACP MF @ Day 14 | DACP MF @ Day 30 | FDP @ Dispense | FDP @ Day 3 | FDP @ Day 14 | FDP @ Day 30
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 26 | 26 | 26 | 26
participants
  20/15 | 5 | 4 | 4 | 2 | 0 | 0 | 1 | 2
  20/20 | 40 | 38 | 40 | 42 | 22 | 24 | 21 | 19
  20/25 | 5 | 8 | 6 | 6 | 4 | 1 | 4 | 5
  20/30 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Binocular Snellen Visual Acuity (VA) at Near (40cm) With Study Lenses
Description: Visual Acuity was tested while reading charts at a distance of 40 cm from the participant with both eyes together. The Snellen fraction 20/20 represents 'normal' near vision. A larger denominator indicates a lower visual acuity.
Time Frame: Up to Day 30
Population: This reporting group includes all randomized and dispensed participants who completed the study.
Measure: Number; unit: participants
Arm/Group | DACP MF @ Dispense | DACP MF @ Day 3 | DACP MF @ Day 14 | DACP MF @ Day 30 | FDP @ Dispense | FDP @ Day 3 | FDP @ Day 14 | FDP @ Day 30
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 26 | 26 | 26 | 26
participants
  20/10 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
  20/12.5 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
  20/16 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0
  20/20 | 19 | 18 | 15 | 23 | 3 | 5 | 5 | 8
  20/25 | 21 | 24 | 25 | 20 | 14 | 10 | 10 | 14
  20/30 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  20/32 | 6 | 6 | 6 | 7 | 7 | 8 | 5 | 4
  20/40 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  20/50 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign in subjects, users, or other persons, whether or not related to the medical device. AEs were collected for the duration of the study (2 months).
Description: AEs were obtained as solicited comments and as observations by the study Investigator as outlined in the study protocol. This analysis population includes all randomized participants who were dispensed study product (79).
Arm/Group | DAILIES® AquaComfort Plus® Multifocal | Focus® DAILIES® Progressives
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/27
Other Adverse Events (participants affected / at risk) | 0/52 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.